CLINICAL TRIAL: NCT05175508
Title: Azacitidine in Combination With or Without All-trans Retinoic Acid in Newly Diagnosed Unfit Acute Myeloid Leukemia or Intermediate,High or Very High Risk Myelodysplastic Syndromes (MDS) as Per IPSS-R Criteria
Brief Title: Aza With or Without ATRA in Newly Diagnosed Unfit AML or Intermediate,High or Very High Risk MDS
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital of Soochow University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SOOCHOW-HY-2021-03
Record Dates: First submitted 2021-11-01; First posted 2022-01-03 (Actual); Last update posted 2022-01-03 (Actual); Status verified 2021-04

CONDITIONS: AML; MDS; Old Age; Debility; Hematologic Cancer
Keywords: acute myeloid leukemia; myelodysplastic syndromes; all-trans retinoic acid; azacitidine
MeSH Terms: conditions — Frailty; Hematologic Neoplasms; Leukemia, Myeloid, Acute; Myelodysplastic Syndromes | interventions — Azacitidine; Tretinoin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Azacytidine Combined With ARTA (Experimental): Azacytidine 75mg/m2/d by IV on days 1-7 of every cycle with ATRA 20mg tid by po on days 1-21 of every cycle 28 days
  Interventions: Drug: Azacitidine; Drug: all trans retinoic acid
- Azacytidine (Experimental): Azacytidine 75mg/m2/d by IV on days 1-7 of every cycle
  Interventions: Drug: Azacitidine

INTERVENTIONS:
Drug: Azacitidine — Azacytidine 75mg/m2/d by IV on days 1-7 of every cycle 28 days
  Other Names: AZA
Drug: all trans retinoic acid — ATRA 20mg tid by po on days 1-21 of every cycle 28 days
  Other Names: ATRA
  Arms: Azacytidine Combined With ARTA

SUMMARY:
This is a randomized, open-label, multicenter study to compare the efficacy and safety of AZA with or without ATRA in newly diagnosed unfit AML or Intermediate,High or Very High Risk MDS

DETAILED DESCRIPTION:
Newly diagnosed unfit AML and Intermediate,High or Very High Risk Myelodysplastic Syndromes (MDS) as Per IPSS-R Criteria are unable to tolerate the intensive chemo-therapy regimens due to their old age and poor physical condition, resulting in limited overall survival. Nowadays, AZA are recommended for unfit acute myeloid leukemia or myelodysplastic syndromes patients with remission rate of 30%~34%. AZA with or without all-trans retinoic acid (ATRA) can cooperatively inhibit leukemia cell proliferation , induce apoptosis and differentiation.

ELIGIBILITY:
Inclusion Criteria:

* Chinese guidelines for the diagnosis and treatment of acute myeloid leukemia (2017 edition)，excludes acute promyelocytic leukemia (M3、APL) and myelodysplastic syndromes(2017 edition)
* Be at least 18 years of age on day of signing informed consent
* Not suitable for newly diagnosed patients with intensive chemotherapy
* Not suitable for newly diagnosed patients with receiving hematopoietic stem cell transplantation
* The proportion of blast cells was below 50% in bone marrow
* Total white blood cell (WBC) count ≤10,000/µL；Must be able to swallow tablets

Exclusion Criteria:

* Malignant neoplasms with other progression
* Serious mental illness uncooperative
* Refusal to join the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2021-05-01 (Actual); Primary Completion 2022-05-01 (Estimated); Study Completion 2023-05-01 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate （ORR) | 6 months
  Number of participants (responders) achieving ORR after the 6 cycle treatments，Overall response rate (ORR) based on the International Working Group (IWG)-2006 criteria, which include complete remission (CR), partial remission (PR), and major hematologic improvement (HI).
Overall survival (OS) | 24months
  time from randomization to death from any cause, or last known date to be alive.
Progression-free survival (PFS) | 24 months
  Progression-free survival (PFS) will be measured from time of enrolling in the clinical trial to the date on which disease progresses or the date on which the patient dies, whichever comes first.

SECONDARY OUTCOMES:
Percentage of Participants Achieving Transfusion Independence (TI) Who are Transfusion Dependent at Baseline | 6 months
  TI is when the participants who were transfusion dependent on RBC and/or Platelet at baseline achieve transfusion independence post baseline. TI is a period of at least 56 days with no transfusion after the date of the first dose of study drug to the last dose of study drug + 30 days, the initiation of post-treatment therapy, or death, whichever is earliest.
Incidence of systemic infections | 6 months
  Incidence of systemic infections

CONTACTS AND LOCATIONS:
Overall Officials: Han Yue, Ph.D, Principal Investigator — The First Affiliated Hospital of Soochow University
Locations (1):
- The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chinese Society of Hematology, Chinese Medical Association. [Chinese guidelines for diagnosis and treatment of myelodysplastic syndromes (2019)]. Zhonghua Xue Ye Xue Za Zhi. 2019 Feb 14;40(2):89-97. doi: 10.3760/cma.j.issn.0253-2727.2019.02.001. No abstract available. Chinese. PMID 30831622
- [Background] Leukemia & Lymphoma Group, Chinese Society of Hematology, Chinese Medical Association. [Chinese guidelines for diagnosis and treatment of adult acute myeloid leukemia (not APL) (2017)]. Zhonghua Xue Ye Xue Za Zhi. 2017 Mar 14;38(3):177-182. doi: 10.3760/cma.j.issn.0253-2727.2017.03.001. No abstract available. Chinese. PMID 28395438
- [Background] Dombret H, Seymour JF, Butrym A, Wierzbowska A, Selleslag D, Jang JH, Kumar R, Cavenagh J, Schuh AC, Candoni A, Recher C, Sandhu I, Bernal del Castillo T, Al-Ali HK, Martinelli G, Falantes J, Noppeney R, Stone RM, Minden MD, McIntyre H, Songer S, Lucy LM, Beach CL, Dohner H. International phase 3 study of azacitidine vs conventional care regimens in older patients with newly diagnosed AML with >30% blasts. Blood. 2015 Jul 16;126(3):291-9. doi: 10.1182/blood-2015-01-621664. Epub 2015 May 18. PMID 25987659
- [Background] Delia M, Carluccio P, Buquicchio C, Vergine C, Greco G, Amurri B, Melpignano A, Melillo L, Cascavilla N, Guarini A, Capalbo S, Tarantini G, Mazza P, Pavone V, Di Renzo N, Specchia G. Azacitidine in the treatment of older patients affected by acute myeloid leukemia: A report by the Rete Ematologica Pugliese (REP). Leuk Res. 2015 Aug 20:S0145-2126(15)30358-1. doi: 10.1016/j.leukres.2015.08.005. Online ahead of print. PMID 26364798
- [Background] Fenaux P, Mufti GJ, Hellstrom-Lindberg E, Santini V, Finelli C, Giagounidis A, Schoch R, Gattermann N, Sanz G, List A, Gore SD, Seymour JF, Bennett JM, Byrd J, Backstrom J, Zimmerman L, McKenzie D, Beach C, Silverman LR; International Vidaza High-Risk MDS Survival Study Group. Efficacy of azacitidine compared with that of conventional care regimens in the treatment of higher-risk myelodysplastic syndromes: a randomised, open-label, phase III study. Lancet Oncol. 2009 Mar;10(3):223-32. doi: 10.1016/S1470-2045(09)70003-8. Epub 2009 Feb 21. PMID 19230772
- [Background] Pappa V, Anagnostopoulos A, Bouronikou E, Briasoulis E, Kotsianidis I, Pagoni M, Zikos P, Tsionos K, Viniou N, Meletis J, Papadaki H, Kioumi A, Galanopoulos A, Vervessou EC, Poulakidas E, Karmas P, Karvounis K, Symeonidis A. A retrospective study of azacitidine treatment in patients with intermediate-2 or high risk myelodysplastic syndromes in a real-world clinical setting in Greece. Int J Hematol. 2017 Feb;105(2):184-195. doi: 10.1007/s12185-016-2115-y. Epub 2016 Nov 4. PMID 27815858
- [Background] Xiang L, Zhou J, Gu W, Wang R, Wei J, Qiu G, Cen J, Xie X, Chen Z. Changes in expression of WT1 during induced differentiation of the acute myeloid leukemia cell lines by treatment with 5-aza-2'-deoxycytidine and all-trans retinoic acid. Oncol Lett. 2016 Feb;11(2):1521-1526. doi: 10.3892/ol.2015.4052. Epub 2015 Dec 23. PMID 26893773
- [Background] Xiang L, Wang R, Wei J, Qiu G, Cen J, Hu S, Xie X, Chen Z, Gu W. Retinoic acid receptor-beta gene reexpression and biological activity in SHI-1 cells after combined treatment with 5-aza-2'-deoxycytidine and all-trans retinoic acid. Acta Haematol. 2015;133(3):279-86. doi: 10.1159/000367586. Epub 2014 Nov 20. PMID 25413479
- [Background] Xiang L, Dong W, Wang R, Wei J, Qiu G, Cen J, Chen Z, Zheng X, Hu S, Xie X, Cao X, Gu W. All-trans retinoic acid enhances the effect of 5-aza-2'-deoxycytidine on p16INK4a demethylation, and the two drugs synergistically activate retinoic acid receptor beta gene expression in the human erythroleukemia K562 cell line. Oncol Lett. 2014 Jul;8(1):117-122. doi: 10.3892/ol.2014.2133. Epub 2014 May 12. PMID 24959230
- [Background] Wu W, Lin Y, Xiang L, Dong W, Hua X, Ling Y, Li H, Yan F, Xie X, Gu W. Low-dose decitabine plus all-trans retinoic acid in patients with myeloid neoplasms ineligible for intensive chemotherapy. Ann Hematol. 2016 Jun;95(7):1051-7. doi: 10.1007/s00277-016-2681-3. Epub 2016 Apr 26. PMID 27116384
- [Background] Lubbert M, Grishina O, Schmoor C, Schlenk RF, Jost E, Crysandt M, Heuser M, Thol F, Salih HR, Schittenhelm MM, Germing U, Kuendgen A, Gotze KS, Lindemann HW, Muller-Tidow C, Heil G, Scholl S, Bug G, Schwaenen C, Giagounidis A, Neubauer A, Krauter J, Brugger W, De Wit M, Wasch R, Becker H, May AM, Duyster J, Dohner K, Ganser A, Hackanson B, Dohner H; DECIDER Study Team. Valproate and Retinoic Acid in Combination With Decitabine in Elderly Nonfit Patients With Acute Myeloid Leukemia: Results of a Multicenter, Randomized, 2 x 2, Phase II Trial. J Clin Oncol. 2020 Jan 20;38(3):257-270. doi: 10.1200/JCO.19.01053. Epub 2019 Dec 3. PMID 31794324

DOCUMENTS (1):
  • Study Protocol (2021-12-22): https://cdn.clinicaltrials.gov/large-docs/08/NCT05175508/Prot_000.pdf